CLINICAL TRIAL: NCT01852812
Title: A Phase III, Open-Label Clinical Trial to Study the Safety and Pharmacokinetics of MK-0476 in Japanese Pediatric Subjects Aged 1 to 15 Years Old With Perennial Allergic Rhinitis
Brief Title: Study of the Safety and Pharmacokinetics of Montelukast (MK-0476) in the Treatment of Japanese Pediatric Participants With Perennial Allergic Rhinitis (MK-0476-520)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0476-520; 132233 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2013-05-09; First posted 2013-05-14 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2022-02

CONDITIONS: Perennial Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Montelukast 4 mg OG/1-5 year olds (Experimental): Participants receive montelukast 4 mg OG in one sachet orally (PO) once daily (QD) at bed time for 4 weeks with an option to continue for an additional 8 weeks (12 weeks total)
  Interventions: Drug: Montelukast Oral Granules (OG)
- Montelukast 5 mg CT/6-9 year olds (Experimental): Participants receive montelukast 5 mg CT in one tablet PO QD at bed time for 12 weeks
  Interventions: Drug: Montelukast Chewable Tablets (CT)
- Montelukast 5 mg CT/10-15 year olds (Experimental): Participants receive montelukast 5 mg CT in one tablet PO QD at bed time for 12 weeks
  Interventions: Drug: Montelukast Chewable Tablets (CT)

INTERVENTIONS:
Drug: Montelukast Oral Granules (OG) — Montelukast 4 mg in one sachet
  Arms: Montelukast 4 mg OG/1-5 year olds
Drug: Montelukast Chewable Tablets (CT) — Montelukast 5 mg in one tablet
  Arms: Montelukast 5 mg CT/10-15 year olds; Montelukast 5 mg CT/6-9 year olds

SUMMARY:
This study will evaluate the safety and pharmacokinetics of montelukast (MK-0476) in the treatment of Japanese pediatric participants with perennial allergic rhinitis (PAR). The primary hypothesis of this study is that montelukast oral granules (OG) and chewable tablets (CT) provide appropriate exposure to montelukast in Japanese pediatric participants with PAR.

ELIGIBILITY:
Inclusion Criteria:

* Weight ≥8 kg
* Diagnosis of PAR and has symptoms of PAR at Visit 1

Exclusion Criteria:

* Past or present medical history of asthma
* Diagosis of acute rhinitis, simple rhinitis, rhinitis congestive, rhinitis atrophic, sinusitis with purulent nasal discharge, rhinitis medicamentosa or nonallergic rhinitis (e.g. vasomotor rhinitis, eosinophilic rhinitis)
* Started hyposensitization therapy or non-specific immunotherapy within 6 months prior to Visit 1
* Medical history of inferior concha mucosal resection, submucous resection of inferior turbinates or other surgery aimed at reduction and/or modulation of nasal mucosa (including electrocoagulation, cryoextraction or application of trichloroacetic acid)
* Clinically significant, active disease of the cardiovascular or hematologic systems or uncontrolled hypertension (1 to 5 year olds: >120/70 mmHg; 6 to 9 year olds: >130/80 mmHg; 10 to 15 year olds: >140/85 mmHg)
* Medical history of stunted growth
* Serious drug allergy
* Treated with other clinical study drug within 3 months prior to Visit 1

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2013-06-07 (Actual); Primary Completion 2013-12-24 (Actual); Study Completion 2013-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Okubo K, Inoue Y, Numaguchi H, Tanaka K, Saito I, Oshima N, Matsumoto Y, Prohn M, Mehta A, Nishida C, Philip G. Montelukast in the treatment of perennial allergic rhinitis in paediatric Japanese patients; an open-label clinical trial. J Drug Assess. 2016 Sep 19;5(1):6-14. doi: 10.1080/21556660.2016.1209507. eCollection 2016. PMID 27785374
- [Derived] Hashiguchi K, Okubo K, Inoue Y, Numaguchi H, Tanaka K, Oshima N, Mehta A, Nishida C, Saito I, Philip G. Evaluation of Montelukast for the Treatment of Children With Japanese Cedar Pollinosis Using an Artificial Exposure Chamber (OHIO Chamber). Allergy Rhinol (Providence). 2018 Jul 13;9:2152656718783599. doi: 10.1177/2152656718783599. eCollection 2018 Jan-Dec. PMID 30027002

RESULTS

PARTICIPANT FLOW:
Groups:
- Montelukast 4 mg OG/1-5 Year Olds: Participants receive montelukast 4 mg oral granules (OG) in one sachet orally (PO) once daily (QD) at bed time for 4 weeks with an option to continue for an additional 8 weeks (12 weeks total)
- Montelukast 5 mg CT/6-9 Year Olds: Participants receive montelukast 5 mg chewable tablets (CT) in one tablet PO QD at bed time for 12 weeks
Period: Overall Study
Arm/Group | Montelukast 4 mg OG/1-5 Year Olds | Montelukast 5 mg CT/6-9 Year Olds | Montelukast 5 mg CT/10-15 Year Olds
Started | 51 | 18 | 18
Completed | 51 | 17 | 17
Not Completed | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Non-compliance With Study Drug | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Montelukast 4 mg OG/1-5 Year Olds: Participants receive montelukast 4 mg OG in one sachet PO QD at bed time for 4 weeks with an option to continue for an additional 8 weeks (12 weeks total)
- Total: Total of all reporting groups
Arm/Group | Montelukast 4 mg OG/1-5 Year Olds | Montelukast 5 mg CT/6-9 Year Olds | Montelukast 5 mg CT/10-15 Year Olds | Total
Number analyzed (Participants) | 51 | 18 | 18 | 87
Age, Continuous [Mean (Standard Deviation); unit: Years] | 3.61 (1.4) | 7.78 (1.3) | 11.3 (1.0) | 6.07 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 8 | 5 | 37
  Male | 27 | 10 | 13 | 50

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experience at Least One Adverse Event (AE)
Description: An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of study drug or protocol-specified procedure, whether or not considered related to the study drug or protocol-specified procedure. Any worsening of a pre-existing condition that is temporally associated with the use of study drug is also an AE. Participants were monitored for the occurrence of AEs for up to 14 days after last dose of study drug (up to a total of 14 weeks). AEs were reported based on the dose of study drug participants received.
Time Frame: Up to 14 days after last dose of study drug (Up to 14 weeks)
Population: The All Subjects as Treated (ASaT) population consisted of all participants who received at least one dose of study drug. Data from the two montelukast 5 mg CT groups (6-9 year olds and 10-15 year olds) were pooled for safety analyses.
Measure: Number; unit: Percentage of participants
Groups:
- Montelukast 5 mg CT/6-15 Year Olds: Participants receive montelukast 5 mg CT in one tablet PO QD at bed time for 12 weeks
Arm/Group | Montelukast 4 mg OG/1-5 Year Olds | Montelukast 5 mg CT/6-15 Year Olds
Number analyzed (Participants) | 51 | 36
Percentage of participants | 74.5 | 55.6

2. Primary Outcome: Percentage of Participants Who Discontinue Study Drug Due to an AE
Description: An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of study drug or protocol-specified procedure, whether or not considered related to the study drug or protocol-specified procedure. Any worsening of a pre-existing condition that is temporally associated with the use of study drug is also an AE. Discontinuations due to an AE were reported based on the dose of study drug participants received.
Time Frame: Up to 12 weeks
Population: The ASaT population consisted of all participants who received at least one dose of study drug. Data from the two montelukast 5 mg CT groups (6-9 year olds and 10-15 year olds) were pooled for safety analyses.
Measure: Number; unit: Percentage of participants
Arm/Group | Montelukast 4 mg OG/1-5 Year Olds | Montelukast 5 mg CT/6-15 Year Olds
Number analyzed (Participants) | 51 | 36
Percentage of participants | 0.0 | 2.8

3. Primary Outcome: Area Under the Time-Concentration Curve (AUC 0-∞) of Montelukast CT and Montelukast OG
Description: Blood samples for pharmacokinetic (PK) assessments were collected at either 1 hour (h) or 3 h post-dose on Day 1 and at either 14 h or 22 h post-dose on Day 28.
Time Frame: Up to Day 28 after first dose of study drug
Population: The All Subjects Pharmacokinetically Evaluable (ASPE) population consisted of all participants from the ASaT population who had an evaluable assessement for this PK parameter and did not have any protocol violation which would interfere with this PK parameter. Data for PK assessments were reported by dose of study drug received and age group.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Montelukast 4 mg OG/1-5 Year Olds | Montelukast 5 mg CT/6-9 Year Olds | Montelukast 5 mg CT/10-15 Year Olds
Number analyzed (Participants) | 51 | 18 | 18
h*ng/mL | 4300 (800) | 4350 (760) | 3500 (620)

4. Primary Outcome: Maximum Plasma Concentration (Cmax) of Montelukast CT and Montelukast OG
Description: Blood samples for PK assessments were collected at either 1 h or 3 h post-dose on Day 1 and at either 14 h or 22 h post-dose on Day 28.
Time Frame: Up to Day 28 after first dose of study drug
Population: The ASPE population consisted of all participants from the ASaT population who had an evaluable assessement for this PK parameter and did not have any protocol violation which would interfere with this PK parameter. Data for PK assessments were reported by dose of study drug received and age group.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Montelukast 4 mg OG/1-5 Year Olds | Montelukast 5 mg CT/6-9 Year Olds | Montelukast 5 mg CT/10-15 Year Olds
Number analyzed (Participants) | 51 | 18 | 18
ng/mL | 510 (84) | 438 (82) | 344 (61)

5. Primary Outcome: Time to Cmax (Tmax) of Montelukast CT and Montelukast OG
Description: as for outcome 4
Time Frame: Up to Day 28 after first dose of study drug
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Montelukast 4 mg OG/1-5 Year Olds | Montelukast 5 mg CT/6-9 Year Olds | Montelukast 5 mg CT/10-15 Year Olds
Number analyzed (Participants) | 51 | 18 | 18
Hours | 2.74 (0.60) | 3.55 (0.71) | 3.65 (0.60)

6. Primary Outcome: Apparent Elimination Half-life (t1/2) of Montelukast CT and Montelukast OG
Description: as for outcome 4
Time Frame: Up to Day 28 after first dose of study drug
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Montelukast 4 mg OG/1-5 Year Olds | Montelukast 5 mg CT/6-9 Year Olds | Montelukast 5 mg CT/10-15 Year Olds
Number analyzed (Participants) | 51 | 18 | 18
Hours | 1.27 (0.56) | 2.01 (0.75) | 2.08 (0.66)

ADVERSE EVENTS:
Time Frame: Up to 14 days after last dose of study drug (Up to 14 weeks)
Description: The ASaT population consisted of all participants who received at least one dose of study drug. AEs were reported based on the dose of study drug participants received. Data from the two montelukast 5 mg CT groups (6-9 year olds and 10-15 year olds) were pooled for safety analyses.
Arm/Group | Montelukast 4 mg OG/1-5 Year Olds | Montelukast 5 mg CT/6-15 Year Olds
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/36
Other Adverse Events (participants affected / at risk) | 37/51 | 18/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Montelukast 4 mg OG/1-5 Year Olds (N=51) | Montelukast 5 mg CT/6-15 Year Olds (N=36)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Acute sinusitis (Infections and infestations) | 6 (8) | 0 (0)
Bronchitis (Infections and infestations) | 3 (4) | 3 (3)
Gastroenteritis (Infections and infestations) | 3 (3) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 22 (32) | 12 (15)
Otitis media (Infections and infestations) | 4 (4) | 1 (1)
Otitis media acute (Infections and infestations) | 3 (4) | 0 (0)
Pharyngitis (Infections and infestations) | 9 (14) | 3 (4)
Arthropod sting (Injury, poisoning and procedural complications) | 2 (2) | 2 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.